CLINICAL TRIAL: NCT00159731
Title: An Open Label Extension Safety Trial of Pregabalin (CI-1008) in Subjects With Diabetic Peripheral Neuropathy
Brief Title: Safety of Pregabalin in the Treatment of Pain Due to Diabetic Peripheral Neuropathy
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Pfizer's Upjohn has merged with Mylan to form Viatris Inc. (Industry)
Responsible Party: Sponsor
Organization: Pfizer (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: A0081036
Record Dates: First submitted 2005-09-08; First posted 2005-09-12 (Estimated); Last update posted 2021-01-22 (Actual); Status verified 2006-07

CONDITIONS: Diabetic Peripheral Neuropathy
MeSH Terms: interventions — Pregabalin

INTERVENTIONS:
Drug: Pregabalin

SUMMARY:
The purpose of this study is to 1) provide continued pregabalin treatment for 6 additional months to patients who have taken part in the placebo controlled study A0081060; and 2) find out if pregabalin is safe at a dose of 600 mg/day (taken twice a day)

ELIGIBILITY:
Inclusion Criteria:

* Adults with Type 1 or 2 diabetes
* Patients must have pain in their lower legs or feet due to painful diabetic neuropathy that has lasted for at least 3 months

Exclusion Criteria:

* Patients must not be in poor or unstable health.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 160
Dates: Start 2005-01; Study Completion 2006-05

PRIMARY OUTCOMES:
Adverse events

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (22):
- United States (22):
  - Pfizer Investigational Site, Hot Springs, Arkansas
  - Pfizer Investigational Site, La Jolla, California
  - Pfizer Investigational Site, Torrance, California
  - Pfizer Investigational Site, Denver, Colorado
  - Pfizer Investigational Site, Ocala, Florida
  - Pfizer Investigational Site, Palm Beach Gardens, Florida
  - Pfizer Investigational Site, Sunrise, Florida
  - Pfizer Investigational Site, West Palm Beach, Florida
  - Pfizer Investigational Site, Boston, Massachusetts
  - Pfizer Investigational Site, Omaha, Nebraska
  - Pfizer Investigational Site, Las Vegas, Nevada
  - Pfizer Investigational Site, Englewood, New Jersey
  - Pfizer Investigational Site, New Brunswick, New Jersey
  - Pfizer Investigational Site, Albany, New York
  - Pfizer Investigational Site, Rochester, New York
  - Pfizer Investigational Site, Greenville, North Carolina
  - Pfizer Investigational Site, Toledo, Ohio
  - Pfizer Investigational Site, Duncansville, Pennsylvania
  - Pfizer Investigational Site, Dallas, Texas
  - Pfizer Investigational Site, Houston, Texas
  - Pfizer Investigational Site, San Antonio, Texas
  - Pfizer Investigational Site, Salt Lake City, Utah

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=A0081036&StudyName=Safety+of+Pregabalin+in+the+Treatment+of+Pain+Due+to+Diabetic+Peripheral+Neuropathy